CLINICAL TRIAL: NCT06430580
Title: Cannabinoids and Biological Reactivity to Stress
Acronym: COBRAS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Wayne State University (Other); National Institute on Drug Abuse (NIDA) (NIH); Auburn University (Other)
Responsible Party: Principal Investigator, Rick James Macatee, Associate Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00006376; R21DA058780-01A1 (NIH)
Record Dates: First submitted 2024-05-13; First posted 2024-05-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Cannabis Use Disorder
MeSH Terms: interventions — Hydrocortisone; Yohimbine

STUDY DESIGN:
Intervention Model Description: 2x2 randomized double-blind within-subject crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 20mg hydrocortisone + 54mg yohimbine hcl (Experimental): 20mg hydrocortisone, single oral dose 54mg yohimbine hcl, single oral dose
  Interventions: Drug: Hydrocortisone Oral; Drug: Yohimbine Hydrochloride
- 20mg hydrocortisone + 54mg placebo (Experimental): 20mg hydrocortisone, single oral dose 54mg cornstarch placebo, single oral dose
  Interventions: Drug: Hydrocortisone Oral; Drug: Cornstarch Placebo 54mg
- 20mg placebo + 54mg yohimbine hcl (Active Comparator): 20mg cornstarch placebo, single oral dose 54mg yohimbine hcl, single oral dose
  Interventions: Drug: Yohimbine Hydrochloride; Drug: Cornstarch Placebo 20mg
- 20mg placebo + 54mg placebo (Placebo Comparator): 20mg cornstarch placebo, single oral dose 54mg cornstarch placebo, single oral dose
  Interventions: Drug: Cornstarch Placebo 20mg; Drug: Cornstarch Placebo 54mg

INTERVENTIONS:
Drug: Hydrocortisone Oral — 20mg hydrocortisone, single oral dose
  Arms: 20mg hydrocortisone + 54mg placebo; 20mg hydrocortisone + 54mg yohimbine hcl
Drug: Yohimbine Hydrochloride — 54mg yohimbine hcl, single oral dose
  Arms: 20mg hydrocortisone + 54mg yohimbine hcl; 20mg placebo + 54mg yohimbine hcl
Drug: Cornstarch Placebo 20mg — 20mg cornstarch placebo, single oral dose
  Arms: 20mg placebo + 54mg placebo; 20mg placebo + 54mg yohimbine hcl
Drug: Cornstarch Placebo 54mg — 54mg cornstarch placebo, single oral dose
  Arms: 20mg hydrocortisone + 54mg placebo; 20mg placebo + 54mg placebo

SUMMARY:
The goal of this study is to test the impact of two drugs that produce temporary stress-like symptoms, both in isolation and together, on cannabis use motivation in individuals with Cannabis Use Disorder. The main questions it will answer are:

1. How do different forms of stress affect cannabis use motivation?
2. How do different forms of stress affect the body's natural cannabinoids?

Researchers will compare a placebo to both drugs in isolation, as well as together, across four separate lab visits.

Participants will:

1) Complete a clinical screening interview (by phone or in-person) and visit the lab for a medical screening, and if eligible:

a) Visit the lab four times where they will: i). Take one of four drug combinations ii). Complete an interview, questionnaires, and computerized tasks iii). Have their brain activity recorded with an EEG cap iv). Provide three blood samples

DETAILED DESCRIPTION:
The prevalence of daily cannabis use and cannabis use disorder (CUD) has increased in the United States over the past two decades. Unfortunately, psychosocial treatments produce minimal long-term abstinence rates and no FDA-approved medications for CUD exist. Thus, identifying novel CUD treatment targets is an increasingly urgent public health need.

Stress-elicited cannabis use motivation has been implicated in worse CUD outcomes, but a mechanistic understanding of how acute stress increases cannabis use motivation in CUD is limited. Prior work has demonstrated that acute psychosocial stress enhancement of subsequent cannabis cue incentive salience, as indexed by the late positive potential (neural measure of approach-motivated attention recorded using electroencephalography [EEG]), was associated with worse CUD severity and intervention response, independent of subjective craving. Moreover, hypothalamic pituitary adrenal [HPA]-axis, rather than noradrenergic or subjective reactivity to the psychosocial stressor was associated with subsequent potentiation of the cannabis cue-elicited late positive potential. These studies suggest that non-genomic, rapid glucocorticoid effects may be a contributing mechanism in stress amplification of neural drug-cue reactivity, but their correlational designs preclude causal inference. Further, psychosocial stressors are unable to isolate HPA-axis vs. noradrenergic components of stress reactivity.

To isolate HPA-axis activation and test causality, pharmacological manipulations, common in animal models but rare in human studies, will be used to produce separate and co-operative glucocorticoid (20mg hydrocortisone) and noradrenergic (54mg yohimbine) activation. The investigators will employ a 2x2 randomized, placebo-controlled double-blind crossover design in 36 participants with severe CUD. The primary aim is to test the causal potentiating effect of glucocorticoids on drug-cue reactivity and drug use motivation, and further determine if the effect depends on co-occurring noradrenergic stimulation. Preclinical work indicates that glucocorticoids can potentiate reward motivation via mobilization of endocannabinoid activity (primary target of cannabis). Thus, as an exploratory aim, the investigators will obtain plasma samples to test the impact of pharmacological stress on circulating endocannabinoids (2-AG, AEA) and their mediating role in glucocorticoid potentiation of drug-cue reactivity and drug use motivation. This project represents a highly novel integration of a rigorous pharmacological challenge design with biological markers of drug-cue incentive salience and endocannabinoid system activity. If hypotheses are confirmed, one causal mechanism through which stress increases neural cannabis cue reactivity will be known, which has immediate implications for testing experimental therapeutics. The long-term goal is to understand how a stress-related mechanism predictive of worse CUD phenotype is generated and can be blocked in CUD. Development of this model will provide a valid, efficient and (relative to other neuroimaging methods) low-cost approach to screen candidate medications and optimize psychosocial drug cue exposure therapies.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for current, moderate to severe Cannabis Use Disorder (CUD) as assessed by the Structured Clinical Interview (SCID) for the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) during the screening interview.
* Reports engagement in near-daily/daily cannabis use.
* Provide a urine sample positive for THC.
* Must be in generally good health as determined by a physical exam, EKG, and blood tests
* Must be adequately informed of the nature and risks of the study and given written informed consent prior to screening.
* Able to read and write in English.

Exclusion Criteria:

* Has a history of serious psychiatric problems (i.e., psychosis, Bipolar Disorder I) or meets criteria for a current Major Depressive Episode, as assessed by the SCID-V-RV.
* Reports current suicidal ideation.
* Meets DSM-5 criteria for any other current, moderate to severe substance use disorder (other than CUD or Tobacco Use Disorder
* Has a positive result urine drug screen for all other drugs aside from THC (i.e., amphetamine, methamphetamine, benzodiazepine, cocaine, MDMA, morphine, oxycodone, methadone, buprenorphine) at screening or at any lab visit.
* Has structural brain abnormalities (e.g., neoplasms), stroke, seizures, infectious disease, a history of other neurological diseases, or a history of head trauma resulting in unconsciousness.
* Has a history of cardiovascular disease, myocardial infarction, chest pain, or palpitations on exertion or drug use, edema, hypertension, resting heart rate <50 BPM or >100 BPM. Cardiovascular diseases include:

  . a. Benign prostatic hyperplasia (BPH) b. Post-myocardial infarction
* Demonstrates systolic BP outside of acceptable range (80-140mmHG), or diastolic BP outside of acceptable range (50-90 mmHG)
* Has a history of cor pulmonale, dyspnea, orthopnea, tachypnea (>24 breaths per minute), or uncontrolled chronic obstructive pulmonary disease or asthma.
* Currently taking any daily psychotropic medication
* Currently taking any of the following medications:

  1. Angiotensin-Converting Enzyme (ACE) inhibitors including Lisinopril, Enalapril, Benazepril, and Bamipril
  2. Angiotensin II Receptor Blockers (ARB) including Losartan, Valsartan, and Olmesartan
  3. Thiazide Diuretics including Hydrochlorothiazide (HCTZ), Chlorthalidone
  4. Calcium Channel Blockers including Amlodipine, Diltiazem, and Verapamil
  5. Beta-blockers including Carvedilol, Metoprolol, Atenolol, Propranolol
  6. Anti-Arrythmic Medication including Disopyramide, Flecainide, and Mexiletine
  7. Edema (Diuretics)
  8. Thiazide Diuretics (as above)
  9. Loop Diuretics including Furosemide and Torsemide
  10. Potassium Sparing Diuretics: Spironolactone and Eplerenone
  11. Anti-Platelet Medications such as Clopidogrel, Prasugrel, and Ticagrelor
* Reproductively capable candidates who are pregnant (based on urine test at screening or at any lab visit) or are heterosexually active and not using medically approved birth control measures (oral contraceptives, IUD, condom, sterilization).
* Self-reports currently seeking or engaging in CUD treatment or any other alcohol or drug treatment.
* Self-reports intent to imminently quit cannabis use.
* Has a Blood-Injection-Injury Phobia, as determined by scores greater than 15 on the Injection and Blood Draw subscale of the Medical Fear Survey

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Amplitude of neurophysiological response to cannabis cues (μV) | Late positive potential amplitude outcome is assessed at each of the four lab visits, which take place over the study period (10-22 days)
  Change in electroencephalography-recorded (EEG) late positive potential amplitude to cannabis cue images after hydrocortisone (with or without yohimbine) compared to placebo+placebo and yohimbine+placebo conditions (higher amplitudes indicate worse outcome)
Amplitude of Demand Intensity for Cannabis (# of hits at $0) | Intensity is assessed at each of the four lab visits, which take place over the study period (10-22 days)
  Marijuana purchase task-derived Intensity after hydrocortisone administration (with or without yohimbine) compared to placebo+placebo and yohimbine+placebo (increased Intensity indicates worse outcome)
Peak Total Monetary Expenditure for Cannabis (total amount of money spent on hits) | OMax is assessed at each of the four lab visits, which take place over the study period (10-22 days)
  Marijuana purchase task-derived OMax after hydrocortisone administration (with or without yohimbine) compared to placebo+placebo and yohimbine+placebo (increased OMax indicates worse outcome)
Breakpoint of Monetary Expenditure for Cannabis (price at which no hits are purchased) | Breakpoint is assessed at each of the four lab visits, which take place over the study period (10-22 days)
  Marijuana purchase task-derived Breakpoint after hydrocortisone administration (with or without yohimbine) compared to placebo+placebo and yohimbine+placebo (increased Breakpoint indicates worse outcome)
Sensitivity of Cannabis Hit Purchasing Behavior to Price Increases | Elasticity is assessed at each of the four lab visits, which take place over the study period (10-22 days)
  Marijuana purchase task-derived Elasticity after hydrocortisone administration (with or without yohimbine) compared to placebo+placebo and yohimbine+placebo (decreased Elasticity indicates worse outcome)
Frequency of implicit cannabis image choice | Implicit choice task # of cannabis image selections outcome is assessed at each of the four lab visits, which take place over the study period (10-22 days)
  Change in cannabis image selections on the Implicit Image Choice Task (computerized behavioral task; range 0-30; higher scores indicate worse outcome) after hydrocortisone administration (with and without yohimbine) compared to placebo+placebo and yohimbine+placebo
Frequency of explicit cannabis image choice | Explicit choice task # of cannabis image selections outcome is assessed at each of the four lab visits, which take place over the study period (10-22 days)
  Change in cannabis image selections on the Explicit Image Choice Task (computerized behavioral task; range 0-30; higher scores indicate worse outcome) after hydrocortisone administration (with and without yohimbine) compared to placebo+placebo and yohimbine+placebo

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Macatee, PhD, Principal Investigator — Florida State University
Locations (1):
- The BRAINS Lab at Florida State University, Tallahassee, Florida, United States